CLINICAL TRIAL: NCT06830824
Title: Effect of Supplementation of a Symbiotic (Inulin + Lactobacillus Acidophilus) on Cognitive Impairment in Older Adults with Type 2 Diabetes Mellitus
Brief Title: Supplementation of Inulin + L. Acidophilus in Elders with T2DM
Status: Not yet recruiting | Phase: Not Applicable | Type: Interventional
Sponsor: Anahuac University (Other)
Responsible Party: Principal Investigator, Jose Juan Antonio Ibarra Arias, Director of Health Research Institute of Universidad Anahuac, Principal Investigator, Anahuac University
Allocation: Randomized | Model: Crossover | Masking: Triple | Purpose: Prevention
Other Study IDs: 202439
Record Dates: First submitted 2025-02-12; First posted 2025-02-17 (Actual); Last update posted 2025-02-19 (Actual); Status verified 2025-02

CONDITIONS: Diabetes Mellitus; Microbiome; Cognition Disorders
Keywords: Diabetes Mellitus; Supplementation; Cognitive impairment
MeSH Terms: conditions — Diabetes Mellitus; Cognition Disorders; Cognitive Dysfunction | interventions — Lacteol

STUDY DESIGN:
Who Masked: Participant, Care Provider, Outcomes Assessor
Oversight: Data Monitoring Committee: Yes | FDA-regulated Drug: No | FDA-regulated Device: No | US Export: No

ARMS (2):
- Phase 1 (Active Comparator)
  Interventions: Dietary Supplement: Lactobacillus acidophilus
- Phase 2 (Placebo Comparator)
  Interventions: Other: Placebo

INTERVENTIONS:
Dietary Supplement: Lactobacillus acidophilus — A pack of symbiotic powder with 1 gram of e. facieum and 8g of agave inulin will be administered daily for 8 weeks
  Arms: Phase 1
Other: Placebo — A pack of unsweetened almond powder milk will be administered daily for 8 weeks
  Arms: Phase 2

SUMMARY:
This study investigates the effects of a symbotic supplement (Inulin + Lactobacillus acidophilus) on cognitive impairment in older adults with type 2 diabetes mellitus (T2DM). Diabetes is a chronic disease characterized by insulin deficiency or resistance, leading to hyperglycemia and long-term complications, including cognitive decline. Cognitive impairment in T2DM patients is linked to oxidative stress, neuroinflammation, and disrupted insulin signaling in the brain.

The gut-brain axis plays a crucial role in cognition, with gut microbiota influencing neuroinflammatory processes. Dysbiosis, common in T2DM, exacerbates cognitive decline. Probiotics like Lactobacillus acidophilus and prebiotics like inulin can restore gut microbiota balance, reduce inflammation, and promote brain-derived neurotrophic factor (BDNF) production, improving cognitive function.

This randomized, crossover clinical trial will enroll 24 patients aged 50-65 with T2DM and mild cognitive impairment. Participants will be divided into control and experimental groups, with an 8-week intervention phase followed by a crossover. The experimental group will receive 8g of inulin and L. acidophilus daily, while the control group will receive a placebo. Cognitive assessments (MMSE, MoCA), PET-CT imaging, gut microbiota sequencing, and butyrate measurements will evaluate the intervention's effects.

The study aims to determine whether symbiotic supplementation can improve cognitive function and metabolic brain activity in T2DM patients. If successful, it may offer an accessible, non-pharmacological approach to mitigating diabetes-related cognitive decline. The research is funded by the Universidad Anáhuac Health Sciences Research Center and international diabetes research organizations.

DETAILED DESCRIPTION:
Study Type: Exploratory with cause and effect direction Study Design: Two-stage, crossover, experimental randomized clinical trial with pretest/posttest. Experiment: Pre-test/post-test design with crossover groups Study population: patients with a diagnosis of type 2 Diabetes, aged 50 to 65 years.

An exploratory study with cause-effect direction will be carried out with an experimental design of randomized clinical trial with crossover pre-test and post-test design. The present protocol is the continuation of a preliminary study with the same characteristics and that upon completion the treated group will become the control group (without treatment) and the control group will become the experimental group (with treatment).

Study population Patients of both sexes from Mexico City and Metropolitan Area with a diagnosis of DM2 with an age range of 50 to 65 years who present mild cognitive disorder, subjected to cognitive function assessment using the Montreal Cognitive Assessment (MoCA) and the Memory Alteration Test (MAT). Recruitment will be carried out by means of promotion in social networks, advertisements posted in clinics and hospitals, as well as contact with general practitioners and/or specialists who may have patients with characteristics matching the study criteria.

Sample size calculation Since this is an exploratory study, it is not necessary to calculate the sample size. However, a minimum of 12 patients is recommended, therefore, in this study it was decided to include a minimum of 12 patients for the control group and 12 for the experimental group. Of the 12 patients, 6 will be women and 6 men for each group.

Phases First Stage (8 weeks of intervention).

* Experimental Group: Will receive symbiotic composed of 8 g of inulin + 1x10 ⁹ CFU of Lactobacillus acidophilus per day for 8 weeks. Control Group: Will consume an almond-based placebo drink for 8 weeks.
* Assessments:
* Cognitive tests (MMSE, MOCA) before and after the intervention. Second Stage (Cross-group, 8 weeks intervention)
* Crossing of Groups:
* The group that was Control in the first stage will become Experimental.
* The group that was Experimental in the first stage will become Control.
* Assessments:
* Cognitive tests (MMSE, MOCA) after 8 weeks of intervention and after 8 weeks of follow-up without treatment.

Final Evaluations

PET-CT with F18-FDG:

* To be performed at the conclusion of both stages using F18-FDG as a marker to analyze brain metabolic changes and evaluate their correlation with cognitive tests.

  2. Stool Microbiota Sequencing:
* Assessment of gut microbiota composition at the end of both stages. 3. Butyrate Measurement:
* Determination of butyrate levels in fecal samples to correlate with cognitive and metabolic outcomes.

Selection Criteria Inclusion criteria Patients between 60-90 years of age with a diagnosis of DM2 who present some degree of cognitive impairment, assessed with the scales. Patients who sign the informed consent form.

Non-inclusion criteria. Related to cognitive impairment, Alzheimer's disease, cerebral ischemia, previous CVE, previous craniocerebral trauma, renal disease grade IIIB or higher. Poor control of systemic arterial hypertension, dyslipidemia and depression diagnosed by DSM V. Patients who do not sign the informed consent C) Exclusion Criteria Patients who in the development of the study present comorbidities that influence cognitive impairment. Patients who present adverse effects to supplementation. Patients who decide to abandon the study or withdraw informed consent. Patients who do not take the symbiotic for 3 consecutive doses.

Instruments for the measurement of the variables Mini-mental (MMSE) It is an instrument for the evaluation of higher mental faculties, specifically it evaluates immediate memory, attention, mathematical calculations and language. It lasts 10 minutes and has a maximum score of 30. The following scores are obtained: Normal (27-30 points): A score of 27 or higher suggests normal cognitive function. However, scores may vary by age and educational level. Mild cognitive impairment (21-26 points): This range indicates mild cognitive impairment, where the person may show some difficulty with cognitive tasks, but is still able to function independently in most daily activities. Moderate cognitive impairment (10-20 points): A score in this range suggests more significant cognitive impairment. The person may have noticeable difficulty with cognitive functions and may need assistance in daily living. Severe cognitive impairment (less than 10 points): A score below 10 indicates severe cognitive impairment, where the person may have significant difficulty performing daily activities and is likely to need constant attention.

Montreal Cognitive Assessment (MOCA) The Montreal Cognitive Assessment is a test designed to assess cognitive impairment. The MoCA has a maximum score of 30 points, and interpretation is based on the following ranges: Normal score (26-30 points): Indicates intact or normal cognitive function. However, it should be noted that this range may vary depending on the age, educational level and language of the individual being assessed. Mild cognitive impairment (18-25 points): Suggests that the person may have mild cognitive difficulties, which may be indicative of initial cognitive impairment. And moderate to severe cognitive impairment (less than 18 points): A score below 18 points indicates moderate to severe cognitive impairment, may be associated with dementia or more advanced cognitive disorders, where the person may have significant difficulties in performing daily tasks.

MoCA is designed to be sensitive in detecting early cognitive deficits, and is useful in the diagnosis of conditions such as Alzheimer's disease and other forms of dementia. As with other cognitive tests, the results should be interpreted in conjunction with other clinical studies and tests, taking into account factors such as the patient's age, educational level, and general health status.

PET-CT with F18-FDG PET-CT with F18-FDG (Fluorine-18-labeled Fluorodeoxyglucose Positron Emission Tomography) is an imaging technique for measuring glucose metabolism in tissues, especially in the brain. F18-FDG is a glucose analog molecule which, when labeled with the radioisotope fluorine-18, emits radiation detectable by the PET scanner.

Principle of Operation

1. Injection of F18-FDG in the patient.
2. Metabolically active cells take up the F18-FDG, especially those that require more glucose (such as neurons).
3. PET detects the radiation emitted by the disintegration of Fluorine-18, generating images showing the distribution of glucose.
4. CT (Computed Tomography) provides detailed anatomical images that are combined with the metabolic data from PET for greater precision.

   Application in Cognitive Impairment

   - Allows the identification of areas of brain hypometabolism associated with cognitive impairment, such as in patients with type 2 diabetes or Alzheimer's disease. Evaluates the effect of therapeutic interventions, such as the use of symbiotics, on brain metabolic activity.

   Advantages - It offers a combined functional and anatomical assessment. -It is a sensitive tool for detecting metabolic changes before structural alterations visible on other imaging techniques appear.

   Within quantitative measurements can be measured:

   SUV (Standardized Uptake Value):

   - Definition: The standard value of glucose uptake in a specific region of the brain.
   * Formula:SUV=Measured activity (MBq/ml)/Injected dose (MBq)/Patient weight (kg)SUV=Injected dose (MBq)/Patient weight (kg)Measured activity (MB q/ml).
   * Normal Range:
   * Normal brain SUV range is usually between 4 and 8 depending on the region and age of the patient.

   CMRglu (Cerebral Metabolic Rate of Glucose):

   - Definition: Measure of the amount of glucose consumed by the brain per unit time.
   * Units: umol/100 g/min.
   * Normal Values: In healthy individuals, it is usually 20-40 umol/100 g/min depending on the brain region.

   Z-Scores:

   - Definition: Scores that compare the F18-FDG uptake of a brain region with reference values.

   - Interpretation:

   - Z > +2: Higher uptake than the reference (hypermetabolism). Z < -2: Lower uptake than the reference (hypometabolism).

   Regions of Interest :

   - Specific areas are evaluated such as:

   - Hippocampus

   - Prefrontal cortex
   * Temporal lobe
   * Parietal lobe Microbiota Sequencing. Microbiota sequencing is a tool to study the composition and function of microorganisms in the human gut. Using DNA sequencing (such as 16S IRNA or shotgun metagenomics), it is possible to analyze the diversity, abundance and functional characteristics of the microorganisms present in the human gut.

     16S rRNA Amplicon Sequencing: The 16S rRNA gene is found in all bacteria and is used to identify bacterial taxa by sequencing the 16S rRNA gene, an specific region of the genome. It is performed quickly, accurately and relatively inexpensively to identify bacterial diversity and determine the microbiological composition of a sample. The limitation is that it can only identify bacteria, not other types of microorganisms such as viruses or fungi.

   Shotgun metagenomics: the shotgun approach sequences all the DNA in a sample (bacteria, viruses, fungi, etc.), providing a more complete view of the microbiota and its potential metabolic functions. Allows for a deeper and more detailed characterization of the microbiota, including metabolic functions and interactions between microorganisms. More expensive and requires more complex bioinformatics analysis Butyrate in feces Gas Chromatography coupled to Mass Spectrometry (GC-MS) GC-MS is one of the most accurate methods for measuring butyrate in feces. This method allows the separation and quantification of volatile fatty acids present in a sample. The procedure consists of the following: Butyrate extraction: fatty acids are extracted from the stool using an organic solvent (e.g., hexane). Derivatization: To improve the volatility of the compounds, the butyrate is converted into a more volatile derivative (e.g. ester). And analysis, the derivative is introduced into a gas chromatograph coupled to a mass spectrometer for separation and quantification. It has a high sensitivity and ability to identify other related metabolites. However; it requires expensive equipment and trained personnel for interpretation of the results.

ELIGIBILITY:
Inclusion Criteria:

* Patients between 60-90 years of age with a diagnosis of DM2 who present some degree of cognitive impairment, assessed with the scales.
* Patients who sign the informed consent form.

Exclusion Criteria:

* Patients who in the development of the study present comorbidities that influence cognitive impairment.
* Patients who present adverse effects to supplementation.
* Patients who decide to abandon the study or withdraw informed consent. - -Patients who do not take the symbiotic for 3 consecutive doses.

Ages: 60 Years to 90 Years | Sex: All | Healthy Volunteers: Yes
Age Groups: Adult, Older Adult
Enrollment: 48 (Estimated)
Dates: Start 2025-03 (Estimated); Primary Completion 2025-08 (Estimated); Study Completion 2025-12 (Estimated)

PRIMARY OUTCOMES:
Cognitive Impairment | 8 weeks
  Change in Score in the Folstein Mini Mental Examination, with a higher score (improvement in cognitive impairment)
  Scoring:
  24-30 Uncertain Cognitive Impairment 18-23 Mild to Moderate Cognitive Impairment 0-17 Severe Cognitive Impairment 0 being the lowest and 30 the highest score obtained
Cognitive Impairment | 8 weeks
  Higher score in Montreal Cognitive Assessment (MoCA), with a total possible score of 30 points, considering a score of 26 or above normal. With the following ranges: Normal range: 26 and above Mild cognitive impairment (MCI): 18-25 Moderate cognitive impairment: 10-17 Severe cognitive impairment: Below 10
Cognitive Impairment | 16 weeks
  PET-CT with F18-FDG:
  To be performed at the conclusion of both stages using F18-FDG as a marker to analyze brain metabolic changes

SECONDARY OUTCOMES:
Stool microbiome | 16 weeks
  Stool Microbiota Sequencing:
  Assessment of gut microbiota composition at the end of both stages
Stool butyrate | 16 weeks
  Butyrate Measurement:
  Determination of butyrate levels in fecal samples to correlate with cognitive and metabolic outcomes.